CLINICAL TRIAL: NCT03196778
Title: Non-Targeted Low Dose Radiotherapy For Recurrent Prostate Cancer
Brief Title: Low Dose Hemi-body Radiation For Recurrent Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juravinski Cancer Center (Other)
Collaborators: McMaster University (Other); Mitacs (Industry); Northern Ontario School of Medicine (Other)
Responsible Party: Principal Investigator, Ian Dayes, Assoc. Professor, Dept of Oncology, Juravinski Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prostate Hemi-body Irradiation
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Dose Radiation (Experimental): Subjects will receive low dose body radiation for 5 weeks.
  Interventions: Radiation: Low Dose Radiotherapy

INTERVENTIONS:
Radiation: Low Dose Radiotherapy — Patients will receive 10 fractions of very low dose hemi-body radiation, delivered, twice per week, over five weeks

SUMMARY:
Older studies in animals and humans have shown cancer responses to very low doses of whole-body or hemi-body radiation. To study the effects of low doses of radiation in patients with recurrent prostate cancer, investigators will enroll up to 21 patients for 10 fractions of low dose radiation, delivered over 5 weeks. Participants will be followed on study for 12 months, capturing PSA, CBC, QoL and blood samples for immunological analysis.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of prostate cancer.
* Having undergone prior prostate surgery or radiotherapy or both.
* Evidence of recurrence of the disease as demonstrated by rising PSA levels. Patients are eligible if on androgen blockade or hormone naïve.

Exclusion Criteria:

* Prior treatment with chemotherapy and/or abiraterone and/or enzalutamide and/or radium-223.
* Receiving treatment with immunosuppressive medications.
* Platelet count below 50,000/µl (50 x 109/l) or leukocyte count below 3,000/µl (3 x 109/l) or granulocyte count below 2,000/µl (2 x 109/l).
* Other medical conditions or co-morbidities which, in the opinion of the Investigator, may interfere with the participant's ability to participate in the study.
* Language difficulties which may hinder the patient's ability to complete the trial.
* Inability of the potential participant to provide consent.
* Lack of independence in daily living activities and any other conditions which, in the opinion of the Investigator, will hinder the participant's ability to participate and complete the study obligations.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
PSA response | Within 12 months of study treatment
  Proportion of patients with a reduction of PSA levels by at least 50%

SECONDARY OUTCOMES:
Immunological changes | Within 12 months of study treatment
  Levels of CD8+ and CD16+ cells, cytokine levels
Adverse Events | Within 12 months of study treatment
  NCI-CTCAE
Quality of Life | Within 12 months of study treatment
  SF-36

CONTACTS AND LOCATIONS:
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD. Results to be reported as aggregate outcomes for the group.

REFERENCES:
- [Derived] Kennedy AE, Dayes IS, Parpia S, Boreham DR, Bowdish DME. Characterizing Hematological Changes Following Repeated Exposure to Non-Targeted Low-Dose Ionizing Radiation in Prostate Cancer Patients. Dose Response. 2024 Oct 2;22(4):15593258241276120. doi: 10.1177/15593258241276120. eCollection 2024 Oct-Dec. PMID 39464181